CLINICAL TRIAL: NCT04685785
Title: Reactibility of Muscle Volume to Ribs Mobilization According to L.Mojzisova.
Brief Title: Reactibility of Muscle Volume to Ribs Mobilization According to Mojžíšová
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Malá Jitka, clinical researcher of physiotherapy department, Charles University, Czech Republic
Other Study IDs: Hofman, Mojzisova
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2020-12

CONDITIONS: Muscle Hypertonia; Rib Syndrome
Keywords: muscle tone, ribs, Mojžišová, joint mobilization
MeSH Terms: conditions — Muscle Hypertonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate a top-rated Prague rehabilitation school´s method. Part of Prague rehabilitation school is called Mojžíšová Method, which is mainly used for the treatment of back pain and woman´s non-structural sterility. This method offers an original, innovative way, how to mobilize 1.- 7. costo-sternal joints. This type of mobilization is very effective, fast and safe and probably widely used only in the Czech Republic. Mojžíšová method uses the excentric force of patients pectoral muscle, passive stretch and shoulder joint internal rotation. According to Mojžíšová, If one of the ribs joints has dysfunction (limited range of motion), there can be found higher sensitivity of this joint, certain muscle reflex spasm, hypersensitive zones and joint dysfunction. Probably the last study evaluating this method was made in the 1990s.

DETAILED DESCRIPTION:
This research aims to analyze the effect of mobilization of 1.-3-ribs joints in a relationship in sensitivity and volume of neck and shoulders muscles. The ultrasonic diagnostic method will be used to evaluate muscle volume before and after mobilization ribs joints. Visual pain scale will be used to evaluate pain during palpation of certain muscles. This research will examine 30 subjects, aged 19-26 years old, which will be divided into the control and the experimental group. Each subject will be in both groups. In the control group, we are going to analyze, if certain neck muscles keep the same volume for 5 minutes during sitting position after ribs mobilization. The control group will evaluate if there are any muscle volume and palpation muscle sensitivity change before and after mobilization of the ribs joints.

Lack of evidence for a relationship between the ribs joints and reflex spasms was the motivation to make this study. During the research, I have found no study, which was aiming to analyze the relationship between the mobilization of ribs joint and reflex muscle spasms.

Subject: Thirty subjects, men and woman, aged from 19 to 26 years old. Each included subject has to be diagnosed with at least one sensitive 1.-3. costo-sternal connection. The study examines the control and the experimental group.

Method: During the entrance diagnostics, the examiner will palpate subject´s 1.-3. costo-sternal connections and certain muscles on the same side of the sensitive connection. Specifically m.scalenus anterior, medius and posterior, sternocleidomastoideus, levator scapulae and trapezius. Those muscles are related to dysfunction of those connections according to Mojžíšová. The subject will rate the sensitivity of those muscles on the visual pain scale (0-10 scale). During palpation, the examiner will be using his index finger. The subject will lay down on their back and turn their head 45 degrees away from the examined side. Then the examiner will use sonograph to evaluate the volume of sternocleidomastoideus, scalenus anterior and medius muscles, on the side, on the side of the sensitive joint. After that, the subject will rest in sitting position for 5 minutes, and then the examiner will use sonograph again to check the volume of those muscles, If there is any volume change without joint mobilization. The subject will be placed in the same position, just as during the first sonographic examination. Those data will be used for the control group.

After this process, the examiner will mobilize 1.-3. costo-vertebral joints, using the Mojžíšová technique. This technique will be done in the sitting position.

ELIGIBILITY:
Inclusion Criteria:

Blockage of first, second and third costovertebral joints and sternocostal distention, hypertension of scalene muscles.

Exclusion Criteria:

Age under 19 and above 26, structural changes and injuries of the cervical spine and upper ribs.

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The observed group composed of University students. Healthy population with typical signs of ribs blockage, according to Mojzisova, means hypertension of surrounded muscles.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Muscle volume changes after joint mobilization | 30 minutes
  Sonography study of muscle volume

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhDr.PhD., Principal Investigator — Faculty of physical education and sport of Charles University
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No